CLINICAL TRIAL: NCT02504905
Title: Propensity to Develop Plasticity in the Parieto-motor Network in Dystonia From the Perspective of Abnormal High-Order Motor Processing
Brief Title: Propensity to Develop Plasticity in the Parieto-Motor Networks in Dystonia From the Perspective of Abnormal High-Order Motor Processing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 150167; 15-N-0167
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Writer's Cramp; Healthy Volunteers; Cervical Dystonia
Keywords: Parietal Lobe; Plasticity; Dystonia; Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Dystonic Disorders; Torticollis; Dystonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAR-CD (Experimental): CD and age/sex matched HV control
  Interventions: Device: TMS
- PAR-WC (Experimental): WC and age/sex matched HV control
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — single TMS pulses at intensities in random order from 0 to 100% (increasing at 5% intervals) of stimulator output at a frequency of 0.1 Hz. Three pulses will be delivered at each intensity. MEPs will be recorded and their amplitudes will be plotted against the corresponding stimulation intensity. This curve will provide three significant parameters: (a) S50 intensity (intensity for which we get a MEP 50 % of its maximal size); (b) estimated resting motor threshold (RMT): the abscissa where the tangent to the slope crosses the x axis; and (c) the maximum MEP ( plateau value).

SUMMARY:
Background:

- People with dystonia have muscle contractions they can t control. These cause slow, repeated motions or abnormal postures. People with dystonia have abnormalities in certain parts of the brain. Researchers want to study the activity of two different brain areas in people with writer s cramp and cervical dystonia.

Objective:

- To compare brain activity in people with dystonia to that in healthy people.

Eligibility:

* Right-handed people ages of 18-65 with cervical dystonia or writer s cramp.
* Healthy volunteers the same ages.

Design:

* Participants will be screened with a physical exam. They will answer questions about being right- or left-handed.
* At study visit 1, participants will:<TAB>
* Have a neurological exam.
* Answer questions about how their disease impacts their daily activities.
* Have a structural magnetic resonance imaging (MRI) scan. Participants will lie on a table that can slide <TAB>in and out of a metal cylinder. This is surrounded by a strong magnetic field.
* Do 2 simple computer tasks.
* At study visit 2:
* Participants will have transcranial magnetic stimulations (TMS) at 2 places on the head. Two wire coils will be held on the scalp. A brief electrical current creates a magnetic pulse that affects brain activity. Muscles of the face, arm, or leg might twitch. Participants may have to tense certain muscles or do simple tasks during TMS. They may be asked to rate any discomfort caused by TMS.
* Muscle activity in the right hand will be recorded by electrodes stuck to the skin of that hand.

DETAILED DESCRIPTION:
Objective:

The purpose of this protocol is to improve understanding of the pathophysiology of dystonia by performing an electrophysiological study using plasticity induction protocols based on dual-site transcranial magnetic stimulation (TMS). We hypothesize that dystonic patients have enhanced responsiveness to plasticity induction in the parieto-motor network. The clinical significance of such an enhanced plasticity will be evaluated by correlating the plasticity measurements with subjects' performance on two tasks engaging high-order motor processing and involving the parietal cortex.

Study population

This study will explore the parieto-motor network (PAR study). There will be two independent arms in each study: one will compare patients with writer s cramp (WC) and age-matched healthy volunteers (HV); and the other one will compare patients with cervical dystonia (CD) with age-matched HVs. The power analysis of thePAR study indicates that we need to enroll 17 patients and 17 healthy volunteers in each arm, with an additional 3 added to account for drop-outs. Therefore, we request a maximum of 20 subjects per patient group and 40 subjects for the control groups.

Design

Subjects will come for one screening visit and two outpatient study visits. During the first study visit patients will be scored clinically for dystonia. They will also undergo a structural magnetic resonance imaging (MRI) to locate the parietal target during the stimulation session. At least 24 hours later, during study visit two, subjects will receive TMS. TMS-induced electromyographic (EMG) activity of hand muscles will be recorded as motor evoked potentials (MEPs). Using single TMS shocks, we will measure at baseline, the input-output (I-O) curve for the right first dorsal interosseous (FDI) muscle MEPs. Then, the subjects will receive a plasticity induction protocol aiming to induce plasticity in the pathway linking the posterior parietal (PP) cortex and the primary motor cortex (M1). To that end, transcranial stimulation will be applied repeatedly (100 pairs) to the left angular gyrus in the PP cortex and to the left M1. At the end of the intervention, the I-O curve will be measured again over the next 50 minutes.

Outcome measures

The amplitude of the MEPs in the I-O curves gives information about corticospinal excitability as a function of TMS stimulation. The primary outcome measure will be the relative change of the MEP size with respect to time (before and 15-20 min after the plasticity intervention). The difference in MEP size will be compared between the HV and the patient groups using a T test.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Between the ages of 18 and 65 years
* Right-handed
* English speaking
* For patients only: confirmed diagnosis of cervical dystonia (PAR-CD) or writer s cramp (PAR-WC).
* For patients treated with anticholinergics and/or benzodiazepines, they must be willing and safely able to abstain from any of these medication for a period of at least 5 plasma half-lives of the individual drug prior to study participation (2 days for trihexyphenidyl which has a plasma half life around 4 hours; 12 days, for clonazepam which has a half-life of 18-50 hours).
* For HVs only: absence of dystonia or other neurological disorder with any effect on the motor or sensory systems
* Ability to give informed consent
* Ability to comply with all study procedures, based on the judgment by the investigator(s).

EXCLUSION CRITERIA:

Any of the following will exclude patients from the study:

* Secondary forms of dystonia, including tardive dyskinesia.
* Dystonic tremor where the tremor is the sole or principal abnormality.
* Botulinum toxin treatment < 3 months prior to visit.

Any of the following will exclude patients or healthy controls from the study:

* Illegal drug use within the past 6 months based on history alone. The intent is to exclude those with drug use that may affect study results.
* Self-reported consumption of 7 alcoholic drinks a week for women and >14 alcoholic drinks a week for man.
* Abnormal findings on neurologic exam (other than dystonia in patient group).
* History of or current brain tumor, stroke, head trauma with loss of consciousness > few seconds, epilepsy or seizures.
* Current diagnosis of major depression or any major mental disorders (axis I disorders).
* Current diagnosis of neurologic disorder other than dystonia.
* Presence of pacemaker, intracardiac lines, implanted pumps or stimulators, or metal objects inside the eye or skull. Dental fillings and dental braces are allowed.
* Known hearing loss.
* Open scalp wounds or scalp infection.
* Current pregnancy.
* Taking benzodiazepines at the time of the study or within 12 days prior to the study.
* Taking anticholinergics at the time of the study or within 2 days prior to the study.
* Taking at the time of the study or within 2 weeks prior to the study any medication that acts as a central nervous system stimulant or that is known to lower seizure threshold, including, imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, foscarnet, ganciclovir, ritonavir, amphetamines, ketamine, gamma-hydroxybutyrate (GHB), theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, antihistamines, and sympathomimetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
MEP size at S50 with respect to time (before, and 15-20 min after PAS intervention) | throughout
  The size of the MEP in the EMG signal gives information about corticospinal excitability as a function of TMS stimulation. An increase in average MEP after the end of PAS intervention implies development of LTP-like plasticity in the pathway linking the parietal cortex or the cerebellum to M1. A decrease would imply development of LTD-like plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Cho, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This protocol pre-dates plans to share IPD, we expect to share deidentified data after publication upon request to comply with NIH policies.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0167.html